CLINICAL TRIAL: NCT07371533
Title: Recombinant Anti-CD19m-CD3 Antibody Injection (A-319) for Refractory/Relapsed or MRD-Positive After Induction Chemotherapy Acute B-Cell Lymphoblastic Leukemia (B-ALL) Clinical Study
Brief Title: Clinical Study of Recombinant Anti-CD19m-CD3 Antibody Injection (A-319)
Acronym: A-319
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM-2025-06
Record Dates: First submitted 2025-11-13; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acute Lymphocytic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1.8 μg/kg dose group (Experimental): The maximum duration of treatment is no more than 4 cycles (one cycle is defined as: 1 week of induction + 3 weeks of treatment + 2 weeks of drug withdrawal). During the 1st week, induction doses of 0.15 μg/kg, 0.45 μg/kg, and 0.9 μg/kg will be administered subcutaneously on Days 1, 3, and 5 respectively. From Weeks 2 to 4, a treatment dose of 1.8 μg/kg will be administered subcutaneously on Days 1, 3, and 5 of each week. Weeks 5 to 6 will be the drug withdrawal period.
  Interventions: Drug: Treatment with A319
- 3.6 μg/kg dose group (Experimental): The maximum duration of treatment is no more than 4 cycles (one cycle is defined as: 1 week of induction + 3 weeks of treatment + 2 weeks of drug withdrawal). During the 1st week, induction doses of 0.15 μg/kg, 0.45 μg/kg, and 0.9 μg/kg will be administered subcutaneously on Days 1, 3, and 5 respectively. From Weeks 2 to 4, a treatment dose of 3.6 μg/kg will be administered subcutaneously on Days 1, 3, and 5 of each week. Weeks 5 to 6 will be the drug withdrawal period.
  Interventions: Drug: Treatment with A319
- 5.0 μg/kg dose group (Experimental): The maximum duration of treatment is no more than 4 cycles (one cycle is defined as: 1 week of induction + 3 weeks of treatment + 2 weeks of drug withdrawal). During the 1st week, induction doses of 0.15 μg/kg, 0.45 μg/kg, and 0.9 μg/kg will be administered subcutaneously on Days 1, 3, and 5 respectively. From Weeks 2 to 4, a treatment dose of 5.0 μg/kg will be administered subcutaneously on Days 1, 3, and 5 of each week. Weeks 5 to 6 will be the drug withdrawal period.
  Interventions: Drug: Treatment with A319

INTERVENTIONS:
Drug: Treatment with A319 — The maximum duration of treatment is no more than 4 cycles (one cycle is defined as: 1 week of induction + 3 weeks of treatment + 2 weeks of drug withdrawal). During the 1st week, induction doses of 0.15 μg/kg, 0.45 μg/kg, and 0.9 μg/kg will be administered subcutaneously on Days 1, 3, and 5 respectively. From Weeks 2 to 4, the corresponding treatment dose will be administered subcutaneously on Days 1, 3, and 5 of each week. Weeks 5 to 6 will be the drug withdrawal period.

SUMMARY:
This is an exploratory study with an open-label, single-arm, single-center design. It plans to enroll subjects with refractory/relapsed acute B-cell lymphoblastic leukemia (B-ALL), or treatment-naive or previously treated B-ALL subjects who achieved complete remission (CR) after induction chemotherapy but still have positive minimal residual disease (MRD). The primary objectives are to preliminarily evaluate the safety, tolerability, pharmacokinetics, biology, preliminary efficacy, and immunogenicity of A-319 subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met for refractory/relapsed acute B-cell lymphoblastic leukemia:

* 1.Aged 18 to 75 years (inclusive), regardless of gender;
* 2.Confirmed diagnosis of refractory or relapsed acute B-cell lymphoblastic leukemia (B-ALL) with positive CD19 expression. Definition of refractory or relapsed: failure to respond to conventional induction chemotherapy; early relapse (relapse within 12 months of first remission); relapse after 12 months of first remission with failure to achieve remission following re-induction with the original regimen; second or subsequent relapse, relapse after autologous hematopoietic stem cell transplantation (Auto-HSCT), or relapse after allogeneic hematopoietic stem cell transplantation (Allo-HSCT). (For patients with Philadelphia chromosome-positive [Ph+] disease, they must have received treatment with at least one tyrosine kinase inhibitor [TKI].);
* 3.Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2;
* 4.Bone marrow blast percentage of at least 5% (determined by morphology);
* 5.Expected life expectancy of at least 3 months;
* 6.Ability to sign the informed consent form and comply with protocol requirements; if the patient is unable to sign, their legal guardian or representative must sign on their behalf.

All of the following criteria must be met for acute B-cell lymphoblastic leukemia (B-ALL) with positive minimal residual disease (MRD) despite achieving complete remission (CR) via induction chemotherapy:

* 1.Aged 18 to 75 years (inclusive), regardless of gender;
* 2.Confirmed diagnosis of acute B-cell lymphoblastic leukemia (B-ALL) with positive CD19 expression;
* 3.B-ALL that has achieved complete morphological remission (CR) via at least 2 cycles of induction chemotherapy# but remains minimal residual disease (MRD)-positive. MRD positivity is defined as detectable nucleated blast cells ≥ 10-⁴. (For patients with Philadelphia chromosome-positive [Ph+] disease, they must have received treatment with tyrosine kinase inhibitors [TKIs] combined with chemotherapy);
* 4.Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 2;
* 5.Ability to sign the informed consent form and comply with protocol requirements; if the patient is unable to sign, their legal guardian or representative must sign on their behalf.

Exclusion Criteria:

* 1.Central nervous system (CNS) leukemia (confirmed by cerebrospinal fluid [CSF] analysis) or acute lymphoblastic leukemia (ALL) with clinically relevant CNS involvement;
* 2.Burkitt's leukemia, testicular infiltration in acute lymphoblastic leukemia (ALL);
* 3.A history of malignancy other than ALL within 5 years prior to the initiation of protocol-specific treatment. Exceptions include: malignancies treated with curative intent, with no known active disease for 5 years before enrollment, and deemed by the treating physician to have a low recurrence risk; non-melanoma skin cancer or lentigo maligna that has been adequately treated with no evidence of recurrence; carcinoma in situ of the cervix that has been adequately treated with no evidence of recurrence; ductal carcinoma in situ of the breast that has been adequately treated with no evidence of recurrence;and prostatic intraepithelial neoplasia with no evidence of prostate cancer;
* 4.Patients with grade 2-4 acute graft-versus-host disease (GVHD) after allogeneic hematopoietic stem cell transplantation (Allo-HSCT), or those with chronic GVHD requiring immunosuppressive therapy;
* 5.Receipt of autologous hematopoietic stem cell transplantation (Auto-HSCT) within 6 weeks, or allogeneic hematopoietic stem cell transplantation (Allo-HSCT) within 3 months, prior to the start of study drug treatment;
* 6.Concurrent chemotherapy, radiotherapy, or systemic treatment for GVHD within 2 weeks prior to the start of study drug treatment;
* 7.Patients with diseases, medical conditions, or social factors that, in the investigator's judgment, may affect study results or compliance. The protocol specifies the following conditions that disqualify patients from participating in the study: uncontrolled acute infection or confirmed bacteremia; known human immunodeficiency virus (HIV) infection, or acute hepatitis B or hepatitis C; patients with severe dyspnea, impaired pulmonary function, or requiring continuous oxygen supplementation; New York Heart Association (NYHA) heart failure classification of grade 3 or 4; myocardial infarction, unstable angina, stroke, transient ischemic attack, severe arrhythmia, or uncontrolled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg) within 6 months prior to drug administration;
* 8.Laboratory test requirements are as follows: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 3 × upper limit of normal (ULN), or > 5 × ULN if liver metastasis is present; total bilirubin > 1.5 × ULN;creatinine clearance < 50 mL/min (calculated using the Cockroft-Gault formula); coagulation function: International Normalized Ratio (INR) > 1.6 (unless on anticoagulant therapy);for patients on oral anticoagulant therapy with a stable dose (for at least 14 days) (e.g., warfarin), INR must be ≤ 3.0 with no bleeding tendency (i.e., no bleeding within 14 days prior to the first dose of the study drug); use of low-molecular-weight heparin is permitted for subjects;
* 9.Previous receipt of anti-CD19 therapy (including CAR-T cell therapy), or immunotherapy (e.g., rituximab) within 4 weeks prior to A-319 treatment;
* 10:Presence of adverse events (except alopecia) caused by anti-tumor treatment that have not resolved to grade 1;
* 11.Pregnant women (positive pregnancy test), lactating women, or women of childbearing potential who refuse to use contraception from the time of signing the informed consent form until at least 3 months after the end of the study; women of childbearing potential must have a positive pregnancy test (human chorionic gonadotropin [HCG] test) within 7 days prior to Day 1 of treatment;
* 12.Male patients (except those who have undergone surgical sterilization) who refuse to use contraception from the time of signing the informed consent form until at least 3 months after the end of the study;
* 13.Known hypersensitivity to the study drug or its excipients;
* 14.Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety Analysis | From the signing of the informed consent form to 30 days after the last dose
  Safety will be evaluated based on the incidence and severity of adverse events (AEs) and serious adverse events (SAEs).
Characteristics of Dose-Limiting Toxicity (DLT) | During the first cycle (each cycle lasts 42 days)
  Dose Limiting Toxicity (DLT) is defined as the occurrence of Grade 3 or higher non-hematologic toxicity (including neurotoxicity) during the first cycle (4 weeks of treatment plus 2 weeks of treatment holiday).

SECONDARY OUTCOMES:
Peripheral Blood Lymphocyte Count | No more than 4 cycles (each cycle is 42 days)
  Pharmacodynamic endpoints:Detection of CD20+, CD19+, CD3+ T cells, CD4+ T cells, and CD8+ T cells.
Maximum Concentration (Cmax) | During the first cycle (each cycle lasts 42 days)
  Pharmacokinetic endpoints
Mean | During the first cycle (each cycle lasts 42 days)
  It will be evaluated based on the levels of cytokines (IL-2, IL-4, IL-6, IL-8, IL-10, IFNγ, TNFα, IL-1β) in peripheral blood.
Best response rate | No more than 4 cycles (each cycle is 42 days)
  Hematologic Complete Remission (CR) or Hematologic Complete Remission with Incomplete Hematologic Recovery (CRi)
Minimal Residual Disease (MRD) Response Rate | No more than 4 cycles (each cycle is 42 days)
Time to Hematologic Relapse | 4 cycles (each cycle is 42 days) plus a 12-month survival follow-up period
  Duration of Response, DOR
Relapse-Free Survival (RFS) | Within 2 years
Overall Survival (OS) | Within 2 years
Percentage of subjects who undergo allogeneic hematopoietic stem cell transplantation (Allo-HSCT) after achieving complete remission (CR), complete remission with incomplete hematologic recovery (CRi), or minimal residual disease (MRD) negativity followi | Within 2 years
Immunogenicity | No more than 4 cycles (each cycle is 42 days)
  Number and percentage of subjects who develop anti-A-319 antibodies (ADA)
Time to Maximum Concentration (Tmax) | During the first cycle (each cycle lasts 42 days)
  Pharmacokinetic endpoints
Area Under the Concentration-Time Curve (AUC) | During the first cycle (each cycle lasts 42 days)
  Pharmacokinetic endpoints
Mean Residence Time (MRT) | During the first cycle (each cycle lasts 42 days)
  Pharmacokinetic endpoints
Apparent Volume of Distribution (Vd) | During the first cycle (each cycle lasts 42 days)
  Pharmacokinetic endpoints
Total Clearance (CL/F) | During the first cycle (each cycle lasts 42 days)
  Pharmacokinetic endpoints
Volume of Distribution (Vz/F) | During the first cycle (each cycle lasts 42 days)
  Pharmacokinetic endpoints
Standard Deviation (SD) | During the first cycle (each cycle lasts 42 days)
  Detection of biomarkers (serum cytokines): Interleukin-2 (IL-2), Interleukin-4 (IL-4), Interleukin-6 (IL-6), Interleukin-8 (IL-8), Interleukin-10 (IL-10), Tumor Necrosis Factor-α (TNF-α), Interferon-γ (IFN-γ), and Interleukin-1β (IL-1β)
Coefficient of Variation (CV) | During the first cycle (each cycle lasts 42 days)
  Detection of biomarkers (serum cytokines): Interleukin-2 (IL-2), Interleukin-4 (IL-4), Interleukin-6 (IL-6), Interleukin-8 (IL-8), Interleukin-10 (IL-10), Tumor Necrosis Factor-α (TNF-α), Interferon-γ (IFN-γ), and Interleukin-1β (IL-1β)

IPD SHARING:
Plan to Share IPD: No